CLINICAL TRIAL: NCT00061256
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of Once-Weekly Alendronate in HIV-Infected Subjects With Decreased Bone Mineral Density Receiving Calcium and Vitamin D
Brief Title: The Effect of Alendronate, Calcium, and Vitamin D on Bone Mineral Density in HIV Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5163; DAIDS-ES ID 10089
Record Dates: First submitted 2003-05-22; First posted 2003-05-23 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections
Keywords: Bone Mineral Density; Lumbar Vertebrae; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Alendronate; Calcium Carbonate; Vitamin D

INTERVENTIONS:
Drug: Alendronate
Drug: Calcium carbonate
Drug: Vitamin D

SUMMARY:
Alendronate is a drug that is used to treat osteoporosis. The purpose of this study is to examine whether alendronate in combination with calcium and vitamin D is safe and effective for treating bone loss in people with HIV.

DETAILED DESCRIPTION:
Decreased bone mineral density (BMD) has been identified in up to 50% of HIV infected men, with severe osteoporosis in up to 21% of these men. The mechanisms underlying these bone abnormalities remain unclear. Bisphosphonates are potent bone resorption inhibitors and have been shown to be effective in treating osteoporosis. While several bisphosphonates are approved for the treatment of osteoporosis in women, alendronate is the only bisphosphonate approved for treatment in men. This study hypothesizes that alendronate will be able to reverse decreased BMD secondary to inhibition of bone resorption in HIV infected patients treated with potent antiretroviral therapy, and that these patients will be able to tolerate alendronate without any significant toxicities. The study will also examine the efficacy of once-weekly alendronate with daily calcium and vitamin D in both men and women with HIV.

Patients will participate in this study for 48 weeks. Patients will be randomly assigned to receive either alendronate or placebo. All patients will receive calcium and vitamin D. Dual energy x-ray absorptiometry (DEXA) scans will be used to evaluate bone density at each visit. After study entry, patients will have visits at Weeks 2, 12, 24, 36, and 48. During these visits, blood will be drawn and a pregnancy test may be performed. Patients must fast for at least 8 hours prior to the entry visit and for the visits at Weeks 2, 12, 24, and 48.

ELIGIBILITY:
Inclusion Criteria

* HIV-1 infection
* Lumbar spine DEXA scan confirming decreased BMD within 90 days prior to study entry
* CD4 cell count 100 cells/mm3 or more within 30 days prior to study entry
* Stable antiretroviral regimen for at least 12 weeks prior to study entry
* No plans to alter antiretroviral therapy or to initiate structured/strategic treatment interruptions
* No plans to significantly alter exercise habits or diet for the duration of the study
* Documentation of two consecutive measurements of viral load of 5000 copies/ml or less within 90 days prior to study entry, with at least one of the two values obtained within 30 days prior to study entry
* Willing to use acceptable methods of contraception
* For women with the absence of menses for at least 6 months, serum prolactin level in the normal range within 60 days prior to study entry
* For women taking estrogen therapy, stable estrogen regimen for at least 24 weeks prior to study entry, with no plan to change estrogen dose for the duration of the study
* Serum calcium between 8 mg/dl and 11 mg/dl within 30 days prior to study entry

Exclusion Criteria

* Men with untreated low total serum testosterone levels within 60 days prior to study entry, or men with plans to initiate testosterone replacement during the study
* Cannot receive vitamin D or calcium supplements
* Daily vitamin or dietary supplements that include 10,000 IU or greater of vitamin A within 90 days prior to study entry
* Hyperparathyroidism, vitamin D deficiency, or oral thrush within 60 days prior to study entry
* Any current or past conditions that predispose to disorders involving the esophagus. Participants with a history of mild or controlled reflux may be enrolled.
* Esophagitis within 6 months prior to study entry
* Pregnant or breastfeeding
* Paget's disease
* Spinal fracture (thoracic or lumbar spine) within 60 days prior to study entry
* Atraumatic bone fracture at any time since 18 years of age
* Spinal fracture at any time in the past
* Inability to stand or sit upright for at least 30 minutes
* Use of systemic glucocorticoids for a cumulative duration of longer than 4 weeks within 6 months immediately prior to study entry
* Use of medications for treatment of osteoporosis within 12 months prior to study entry
* Allergy/hypersensitivity to any component of alendronate, the components of the tablet, or bisphosphonate compounds
* Active drug or alcohol dependence which, in the opinion of the investigator, would interfere with adherence to study requirements or would endanger the patient's health while on study
* Hospitalization for alcohol-related liver disease at any time in the past
* Current use of systemic cytotoxic chemotherapy
* Acute illness within 30 days prior to study entry which, in the opinion of the investigator, would interfere with participation in the study
* History of hepatitis C virus infection
* For participants using anabolic steroids, use of steroids for less than 6 months prior to entry or plans to change current regimen during the course of the study; if a steroid regimen has been discontinued, it must have been discontinued at least 6 months prior to entry

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace McComsey, MD, Study Chair — Division of Infectious Diseases, Case Western Reserve University
Locations (28):
- United States (28):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - UCLA School of Medicine, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - San Francisco General Hospital, San Francisco, California
  - Stanford Univ, Stanford, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Cook County Hospital Core Center, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Univ of Minnesota, Minneapolis, Minnesota
  - Nebraska Health System, Omaha, Nebraska
  - Chelsea Clinic, New York, New York
  - NYU/Bellevue, New York, New York
  - AIDS Community Health Center, Rochester, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hosp, Providence, Rhode Island
  - Stanley Street Treatment and Resource, Providence, Rhode Island
  - The Miriam Hosp, Providence, Rhode Island
  - Comprehensive Care Clinic, Nashville, Tennessee
  - Univ of Texas, Galveston, Galveston, Texas
  - University of Washington (Seattle), Seattle, Washington

REFERENCES:
- [Background] Tebas P, Powderly WG, Claxton S, Marin D, Tantisiriwat W, Teitelbaum SL, Yarasheski KE. Accelerated bone mineral loss in HIV-infected patients receiving potent antiretroviral therapy. AIDS. 2000 Mar 10;14(4):F63-7. doi: 10.1097/00002030-200003100-00005. PMID 10770534
- [Background] Reid IR. The roles of calcium and vitamin D in the prevention of osteoporosis. Endocrinol Metab Clin North Am. 1998 Jun;27(2):389-98. doi: 10.1016/s0889-8529(05)70011-6. PMID 9669144
- [Background] Orwoll E, Ettinger M, Weiss S, Miller P, Kendler D, Graham J, Adami S, Weber K, Lorenc R, Pietschmann P, Vandormael K, Lombardi A. Alendronate for the treatment of osteoporosis in men. N Engl J Med. 2000 Aug 31;343(9):604-10. doi: 10.1056/NEJM200008313430902. PMID 10979796
- [Background] Schnitzer T, Bone HG, Crepaldi G, Adami S, McClung M, Kiel D, Felsenberg D, Recker RR, Tonino RP, Roux C, Pinchera A, Foldes AJ, Greenspan SL, Levine MA, Emkey R, Santora AC 2nd, Kaur A, Thompson DE, Yates J, Orloff JJ. Therapeutic equivalence of alendronate 70 mg once-weekly and alendronate 10 mg daily in the treatment of osteoporosis. Alendronate Once-Weekly Study Group. Aging (Milano). 2000 Feb;12(1):1-12. PMID 10746426
- [Background] Mondy K, Tebas P. Emerging bone problems in patients infected with human immunodeficiency virus. Clin Infect Dis. 2003 Apr 1;36(Suppl 2):S101-5. doi: 10.1086/367566. PMID 12652379
- [Derived] McComsey GA, Kendall MA, Tebas P, Swindells S, Hogg E, Alston-Smith B, Suckow C, Gopalakrishnan G, Benson C, Wohl DA. Alendronate with calcium and vitamin D supplementation is safe and effective for the treatment of decreased bone mineral density in HIV. AIDS. 2007 Nov 30;21(18):2473-82. doi: 10.1097/QAD.0b013e3282ef961d. PMID 18025884
- See also: Click here for more information about alendronate. — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a601011.html
- See also: Click here for more information about calcium carbonate. — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a601032.html